CLINICAL TRIAL: NCT03543956
Title: Professional and Personal Toxic Exposure in Systemic Sclerosis : Type, Intensity and Probability of Exposition
Acronym: VISSEXPOSITION
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/09
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Systemic Sclerosis
Keywords: Silica; Organic Solvents; Toxic substances exposure
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Systemic Sclerosis patient: patients affected by SSc according to EULAR 2013 criteria
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire

SUMMARY:
Systemic Sclerosis (SSc) is an inflammatory chronic disease that can lead to structural damage and handicap. The SSc physiopathology is multifactorial, including genetic and environmental risk factors. The identification of environmental factors implication is crucial to understand the SSc mechanism, and improves the diagnosis and the treatment of the disease.

DETAILED DESCRIPTION:
Studies show that the risk associated with high cumulative exposure to silica and organic solvents appears to be strongly increased in SSc. Moreover, exposure to silica is associated with a specific type of SSc phenotype with a worse prognosis. However, the type, intensity and probability of these expositions are unknown.

The aim of the study is to precisely determine type, intensity and probability of toxic substances exposition in Systemic Sclerosis patients through an auto-questionnaire and integration of these data in a computer matrix.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old
* Speaking and understanding French language
* Being informed about the study and having given his consent
* Affected by SSc according to EULAR 2013 criteria

Exclusion Criteria:

* Patient under tutorship
* Patient who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by SSc according to EULAR 2013 criteria.
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Analyse type, intensity and probability of toxic substances exposition in Systemic Sclerosis patients through an auto-questionnaire and integration of these data in a computer matrix | At baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elise TRUCHETET, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de rhumatologie, Bordeaux, France

REFERENCES:
- [Derived] Galli G, De Pous-Gerardin C, Hanguehard R, Berthy F, Le Moal C, Lourde C, Barnetche T, Skopinski S, Contin-Bordes C, Delva F, Carles C, Truchetet ME. Occupational quantitative exposure to crystalline silica, solvents and pesticides and risk of clinical forms of systemic sclerosis. Rheumatology (Oxford). 2024 Dec 1;63(12):3397-3406. doi: 10.1093/rheumatology/kead602. PMID 37963059